CLINICAL TRIAL: NCT00076388
Title: A Randomized, Open-Label, Parallel Group, International, Multicenter, Phase III Study of Oral ZD1839 (IRESSA®) Versus Intravenous Docetaxel (TAXOTERE®) in Patients With Locally Advanced or Metastatic Recurrent Non-Small Cell Lung Cancer Who Have Previously Received Platinum-Based Chemotherapy
Brief Title: Iressa Versus Docetaxel (Taxotere)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D791GC00001; EudraCT No: 2004-002943-28; 1839IL/0721
Record Dates: First submitted 2004-01-21; First posted 2004-01-23 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Docetaxel

INTERVENTIONS:
Drug: Gefitinib
Drug: Docetaxel

SUMMARY:
The purpose of this study is to compare the effects of ZD1839 or docetaxel in patients with advanced non-small cell lung cancer (NSCLC) that has recurred or progressed after receiving prior treatment with platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Measurable (uni dimensional) disease by RECIST criteria in a lesion not previously irradiated or non measurable disease
* Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy
* Advanced non-small cell lung cancer (NSCLC) that has recurred or progressed after receiving prior treatment with platinum-based chemotherapy
* WHO performance status (PS) 0-2
* Absolute Neutrophil Count (ANC) >1.5 x 109/liter (L) and platelets >100 x 109/L
* Life expectancy of at least 8 weeks

Exclusion Criteria:

* Prior ZD1839 therapy
* Prior docetaxel treatment for NSCLC
* Less than 14 days since completion of prior radiotherapy
* Less than 21 days since prior chemotherapy, immunotherapy or biological systemic anticancer therapy
* Evidence of clinically active Interstitial Lung Disease
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Newly diagnosed CNS metastases that have not yet been treated with surgery and/or radiation. Patients with previously diagnosed and treated CNS metastases or spinal cord compression may be considered if they have evidence of clinically SD (no steroid therapy or steroid dose being tapered) for at least 28 days
* Patients with pre existing peripheral neuropathy >= grade 2 (NCI CTC criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To compare overall survival between ZD1839 and docetaxel

SECONDARY OUTCOMES:
To compare time to progression (TTP) between ZD1839 and docetaxel
To compare progression-free rates at 4 months and 6 months between ZD1839 and docetaxel
To compare the overall objective tumor response rate between ZD1839 and docetaxel
To compare patient-reported functionality (PRF) and quality of life (QoL) between ZD1839 and docetaxel
To compare safety and tolerability of ZD1839 and docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (162):
- United States (35):
  - Research Site, Birmingham, Alabama
  - Research Site, Fountain Valley, California
  - Research Site, Los Angeles, California
  - Research Site, Santa Rosa, California
  - Research Site, Stockton, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Norwich, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Boca Raton, Florida
  - Research Site, Orlando, Florida
  - Research Site, Macon, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Skokie, Illinois
  - Research Site, Knoxville, Kentucky
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Great Neck, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Racine, Wisconsin
- Argentina (8):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research site, El Palomar
  - Research Site, Mar del Plata
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Belgium (8):
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Genk
  - Research Site, Godinne
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Yvoir
- Brazil (3):
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
- Canada (14):
  - Research Site, Edmonton, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Saint Catherines, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, York, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Ste-Foy, Quebec
- China (3):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shanghai
- Croatia (2):
  - Research Site, Split
  - Research Site, Zagreb
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Arhus C
  - Research Site, Glostrup Municipality
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Vejle
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- France (11):
  - Research Site, Blois
  - Research Site, Boulogne-Billancourt
  - Research Site, Caen
  - Research Site, Grenoble
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Nantes
  - Research Site, Niort
  - Research Site, Saint-Herblain
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vesoul
- Germany (17):
  - Research Site, Heidelberg, Baden-Wurttemberg
  - Research Site, Ulm, Baden-Wurttemberg
  - Research Site, Cottbus, Brandenburg
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Bad Segeberg, Schleswig-Holstein
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Großhansdorf
  - Research Site, Leverkusen
  - Research Site, Löwenstein
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Stuttgart
  - Research Site, Wiesbaden
- Research Site, Hong Kong, Hong Kong
- Indonesia (2):
  - Research Site, Jakarta
  - Research Site, Yogyakarta
- Italy (14):
  - Research Site, La Torretta, Ancona
  - Research Site, Bari, BA
  - Research Site, Bergamo, BG
  - Research Site, Bologna, BO
  - Research Site, Cuneo, CN
  - Research Site, Catania, CT
  - Research Site, Forlì, FO
  - Research Site, Melegnano, MI
  - Research Site, Rozzano, MI
  - Research Site, Modena, MO
  - Research Site, Parma, PR
  - Research Site, Roma, Roma
  - Research Site, Torino, TO
  - Research Site, Napoli
- Research Site, Riga, Latvia
- Malaysia (2):
  - Research Site, Kampung Baharu Nilai
  - Research Site, Kuala Lumpur
- Mexico (4):
  - Research Site, Guadalajara
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Torreón
- Philippines (2):
  - Research Site, Manila
  - Research Site, Quezon City
- Research Site, Singapore, Singapore
- Research Site, Ljubliana, Slovenia
- Spain (9):
  - Research Site, Elche, Alicante
  - Research Site, Barcelona, Barcelona
  - Research Site, Girona, Gerona
  - Research Site, Madrid, Madrid
  - Research Site, Málaga, Málaga
  - Research Site, Seville, Sevilla
  - Research Site, Valencia, Valencia
  - Research Site, Vitoria-Gasteiz
  - Research Site, Zaragoza
- Sweden (9):
  - Research Site, Gothenburg
  - Research Site, Luleå
  - Research Site, Örebro
  - Research Site, Östersund
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Umeå
  - Research Site, Västerås
- Switzerland (3):
  - Research Site, Bellinzona
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Research Site, Chiang Mai, Thailand
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir

REFERENCES:
- [Derived] Lombard A, Mistry H, Aarons L, Ogungbenro K. Dose individualisation in oncology using chemotherapy-induced neutropenia: Example of docetaxel in non-small cell lung cancer patients. Br J Clin Pharmacol. 2021 Apr;87(4):2053-2063. doi: 10.1111/bcp.14614. Epub 2020 Dec 19. PMID 33075149
- [Derived] Douillard JY, Shepherd FA, Hirsh V, Mok T, Socinski MA, Gervais R, Liao ML, Bischoff H, Reck M, Sellers MV, Watkins CL, Speake G, Armour AA, Kim ES. Molecular predictors of outcome with gefitinib and docetaxel in previously treated non-small-cell lung cancer: data from the randomized phase III INTEREST trial. J Clin Oncol. 2010 Feb 10;28(5):744-52. doi: 10.1200/JCO.2009.24.3030. Epub 2009 Dec 28. PMID 20038723
- [Derived] Kim ES, Hirsh V, Mok T, Socinski MA, Gervais R, Wu YL, Li LY, Watkins CL, Sellers MV, Lowe ES, Sun Y, Liao ML, Osterlind K, Reck M, Armour AA, Shepherd FA, Lippman SM, Douillard JY. Gefitinib versus docetaxel in previously treated non-small-cell lung cancer (INTEREST): a randomised phase III trial. Lancet. 2008 Nov 22;372(9652):1809-18. doi: 10.1016/S0140-6736(08)61758-4. PMID 19027483